CLINICAL TRIAL: NCT06648070
Title: "Effects of Neuromuscular Reeducation Versus Post Facilitation Stretch Technique for Upper Cross Syndrome Among IT Professionals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/39
Record Dates: First submitted 2024-10-01; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Upper Cross Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMR Group (Experimental): On group A we will perform NEUROMUSCULAR REEDUCATION TECHNIQUE:
  we perform this technique on tight muscles which are:
  1. levator scapulae
  2. upper trapezius
  3. pectoralis major
  Interventions: Procedure: Neuromuscular reeducation technique
- PFS Group (Experimental): On group B we perform POST FACILITATION STRETCH TECHNIQUE on tight muscles same as group A
  1. levator scapulae
  2. upper trapezius
  3. pectoralis major
  Interventions: Procedure: Post Facilitation Stretch

INTERVENTIONS:
Procedure: Neuromuscular reeducation technique — 5 repetitions of neuromuscular reeducation technique i.e. deep pressure along muscles origin to insertion with active movement of that muscle with 10 seconds rest of each repetitions.
  Control group will receive 3- 5 repetitions of Post Facilitation stretch to the tight muscles of UCS i.e. 20% maximal isometric contraction of the muscles to be stretched for 5-10 seconds followed by a rapid stretch ( through the new barrier) of 10 seconds. After stretch muscle is allowed to relax in mid range for 10 seconds.
  Arms: NMR Group
Procedure: Post Facilitation Stretch — 3- 5 repetitions of Post Facilitation stretch to the tight muscles of UCS i.e. 20% maximal isometric contraction of the muscles to be stretched for 5-10 seconds followed by a rapid stretch ( through the new barrier) of 10 seconds. After stretch muscle is allowed to relax in mid range for 10 seconds.
  Arms: PFS Group

SUMMARY:
This study is a randomised control trial and the purpose of this study is to determine the "Effects of Neuromuscular Reeducation Versus Post Facilitation Stretch Technique for Upper Cross Syndrome among IT professionals .

DETAILED DESCRIPTION:
The purpose of this study is to determine the "Effects of Neuromuscular Reeducation Versus Post Facilitation Stretch Technique for Upper Cross Syndrome among IT professionals

we make 2 groups control and treatment group . we give NMR technique to treatment group and PFS technique to control group in patients with upper cross syndrome.

first we take base line readings of cervical ROM , NPRS AND neck diasbilty index.

after 2 weeks of treatment again we take same readings and compare both readings.

with techniques we also perform strengthning excercise of weal muscles for both groups

ELIGIBILITY:
Inclusion Criteria:

* IT profressionals
* 20 - 40 years
* Both genders
* Diagnosed UCS
* Pain from 2 months
* Minimum 4 - 6 hiurs working

Exclusion criteria:

* History of cervical spine
* Fracture
* Trauma to neck

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in ROM | 2 weeks
  ROM will be measured with goniometer
Pain intensity | 2 weeks
  It will be measured using Numeric pain rating scale
Neck Disability | 2 weeks
  It will be measured using Neck disability index

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan